CLINICAL TRIAL: NCT01899261
Title: A Pilot Study of Stereotactic Liver Irradiation for Hepatocellular Carcinoma
Brief Title: Stereotactic Body Radiation Therapy in Treating Patients With Liver Cancer That Cannot Be Removed by Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Nitin Ohri, Principal Investigator, Albert Einstein College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-326; 2010-326 (Other: Albert Einstein College of Medicine); P30CA013330 (NIH)
Record Dates: First submitted 2013-07-11; First posted 2013-07-15 (Estimated); Results first posted 2020-01-22 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Adult Hepatocellular Carcinoma; Advanced Adult Hepatocellular Carcinoma; Localized Non-Resectable Adult Liver Carcinoma; Recurrent Adult Liver Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery

ARMS (1):
- Treatment (SBRT) (Experimental): Patients undergo SBRT every other day over 2 weeks (5 fractions total) in the absence of unacceptable toxicity.
  Interventions: Radiation: Stereotactic Radiosurgery

INTERVENTIONS:
Radiation: Stereotactic Radiosurgery — Undergo SBRT
  Other Names: Stereotactic External Beam Irradiation; stereotactic external-beam radiation therapy; Stereotactic Radiation Therapy; Stereotactic Radiotherapy; stereotaxic radiation therapy; stereotaxic radiosurgery

SUMMARY:
This pilot clinical trial studies stereotactic body radiation therapy in treating patients with liver cancer that cannot be removed by surgery. Stereotactic radiation therapy may be able to send x-rays directly to the tumor and cause less damage to normal tissue.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate feasibility and safety of stereotactic body radiation therapy (SBRT) of the liver for treatment of hepatocellular carcinoma (HCC).

SECONDARY OBJECTIVES:

I. To evaluate radiographic local response, local control and time to local progression (TTLP) of treated lesions in HCC patients after liver SBRT.

II. To evaluate overall survival (OS) and cancer specific survival (CSS) in HCC patients treated with liver SBRT.

III. To evaluate explanted irradiated liver tissue (for patients who proceed to liver transplantation) to determine extent of residual tumor and extent of radiation effects within and around the irradiated field.

OUTLINE:

Patients undergo SBRT every other day over 2 weeks (5 fractions total) in the absence of unacceptable toxicity.

After completion of study treatment, patients are followed up at 1, 3, 6, 9, and 12 months and then every 6 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy > 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* HCC diagnosed by either of the following approaches:

  * Histologic confirmation of HCC on biopsy
  * Evidence of vascular enhancement of suspected lesion on at least two imaging techniques
  * Evidence of vascular enhancement on a single technique if the alpha-fetoprotein (AFP) is > 200 ng/mL in the setting of cirrhosis or chronic hepatitis B/C
* HCC must be deemed unresectable by an experienced surgeon or patient must be medically inoperable or extra-hepatic metastases must be present (making resection an inappropriate treatment option) or patient must have declined the option of surgery after consultation with a surgeon

  * Barcelona Clinic Liver Cancer score of B or C required (i.e., intermediate or advanced stage HCC)
* Prior liver resection or ablative therapy is permitted
* Prior transarterial chemoembolization (TACE) is permitted
* Patients must have recovered from the effects of previous therapy
* Maximal tumor size of 15 cm and > 700 cc of uninvolved liver
* Hemoglobin > 9.0 g/L
* Absolute neutrophil count >= 1.0 bil/L
* Platelets >= 70,000 bil/L
* Total bilirubin < 2 mg/dL
* International normalized ratio (INR) =< 1.5 or correctable with vitamin K (higher INR acceptable if patient is on Coumadin)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) =< 6 times upper range of normal

Exclusion Criteria:

* Active hepatitis or encephalopathy related to liver failure
* Prior radiation therapy to the upper abdomen or thorax
* Lesions within 1 cm from the stomach
* Prior uncontrolled, life threatening malignancy within the previous 6 months
* Pregnancy is not permitted; women of child-bearing age must undergo pregnancy testing prior to enrollment
* Previous gastric, duodenal or variceal bleed within the past 2 months
* Thrombolytic therapy within 4 weeks or commencement of anticoagulant use within the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-10-07 (Actual); Primary Completion 2016-05-09 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Ohri, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (SBRT)
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (SBRT)
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 67 [55 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 6
  More than one race | 5
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 20
Child-Pugh Score [Count of Participants; unit: Participants] — The Child-Pugh score employs five clinical measures of liver disease: total bilirubin, serum albumin, prothrombin time, ascites, and hepatic encephalopathy. Each measure is scored 1-3, with 3 indicating most severe derangement. The total score therefore ranges from 5 to 15.
  Participants
    5 | 10
    6 | 7
    7 | 3

OUTCOME MEASURES:

1. Primary Outcome: Severe Treatment-related Toxicity
Description: The percentage of patients who have severe treatment-related toxicity will be computed, along with exact 95% confidence intervals. Severe toxicity will be defined as grade 4 or 5 hepatic toxicity, thrombocytopenia, or gastrointestinal toxicity, graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0
Time Frame: Within 3 months of SBRT
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (SBRT)
Number analyzed (Participants) | 20
Participants | 0

2. Secondary Outcome: Cancer Specific Survival (CSS)
Description: Cancer Specific Survival (CSS) was assessed in patients who were diagnosed with HCC and treated with liver SBRT as the percentage of patients with Cause-Specific Death from HCC. Patients alive at the end of the follow-up period were censored. Competing risk analysis was performed.
Time Frame: Time from study entry to death from Hepatocellular Carcinoma (HCC) progression, assessed up to 2 years
Measure: Number; unit: percentage of patients
Arm/Group | Treatment (SBRT)
Number analyzed (Participants) | 20
percentage of patients | 10

3. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival, estimated using the Kaplan-Meier method, reflected the percentage of patients who were were diagnosed with HCC and started SBRT treatment and were still alive at the conclusion of the study.
Time Frame: Time from study entry to death from any cause, assessed up to 2 years
Measure: Number; unit: percentage of patients
Arm/Group | Treatment (SBRT)
Number analyzed (Participants) | 20
percentage of patients | 65

4. Secondary Outcome: Time to Local Progression (TTLP) of Treated Lesions
Description: Time to Local progression (TTLP) of treated lesions in HCC patients after liver SBRT treatment was evaluated using Response Evaluation Criteria In Solid Tumors Criteria (RECIST). For patients who died from the study disease without progression of the radiated lesion, time to local progression was censored at the date of death. For patients not known to have died as of the data cut-off date, and who did not have locally progressive disease, time to local progression was censored at the last progression-free disease assessment.
Time Frame: From date of first treatment dose to the first date of objective local progressive disease as defined by RECIST criteria, assessed up to 2 years
Population: 2 subjects with local progression after Stereotactic Body Radiation Therapy (SBRT)
Measure: Mean (Full Range); unit: months
Arm/Group | Treatment (SBRT)
Number analyzed (Participants) | 2
months | 6 [1 to 11]

ADVERSE EVENTS:
Arm/Group | Treatment (SBRT)
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 8/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (SBRT) (N=20)
Fatigue (General disorders) | 3 (3) — Grade 1 fatigue
Nausea (Gastrointestinal disorders) | 2 (2) — Grade 1 nausea
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) — Grade 1 thrombocytopenia
Abdominal pain (Gastrointestinal disorders) | 1 (1) — Grade 1 abdominal pain
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) — Grade 1 dermatitis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes